CLINICAL TRIAL: NCT01121484
Title: A Multicenter, Parallel-Group, Randomized, 10-Week, Double-Blind, Placebo-Controlled Study To Evaluate The Efficacy And Safety Of 50 mg Of DVS SR In The Treatment Of Peri- And Postmenopausal Women With Major Depressive Disorder
Brief Title: Study Evaluating Desvenlafaxine Succinate Sustained-Release (DVS SR) In The Treatment Of Peri- And Postmenopausal Women With Major Depressive Disorder (DVS 3364)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3151A1-3364; B2061029
Record Dates: First submitted 2010-05-03; First posted 2010-05-12 (Estimated); Results first posted 2012-03-30 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-01

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Desvenlafaxine Succinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- desvenlafaxine succinate sustained-release (Experimental)
  Interventions: Drug: desvenlafaxine succinate sustained-release
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: desvenlafaxine succinate sustained-release — 50-mg DVS SR tablets taken orally once daily.
  Other Names: Pristiq
  Arms: desvenlafaxine succinate sustained-release
Drug: placebo — Placebo tablets taken orally once daily.
  Arms: Placebo

SUMMARY:
A multicenter, 10-week study to evaluate the efficacy and safety of 50 mg of desvenlafaxine succinate sustained-release formulation (DVS SR) versus placebo in the treatment of peri- and postmenopausal women with major depressive disorder

ELIGIBILITY:
Inclusion Criteria:

* Peri- and postmenopausal women aged 40 to 70 years who are fluent in both written and spoken English.
* Postmenopausal status defined by 12 consecutive months of spontaneous amenorrhea; less than 12 consecutive months with at least 6 consecutive months of spontaneous amenorrhea and a pre-baseline follicle-stimulating hormone (FSH) level >40 mIU/mL; or 6 months postsurgical bilateral oophorectomy (with or without hysterectomy). Perimenopausal women defined by the presence of any of the following within 6 months before baseline:

  1. an absolute change of 7 days or more in menstrual cycle length within 6 months before baseline;
  2. a change in menstrual flow amount (2 or more flow categories, eg, from light or moderately light to moderately heavy or heavy);
  3. a change in duration (absolute change of 2 or more days); or
  4. periods of amenorrhea lasting at least 3 months.
* A primary diagnosis of major depressive disorder (MDD) based on the criteria in the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition-Text Revision (DSM-IV-TR), single or recurrent episode, without psychotic features using the modified Mini International Neuropsychiatric Interview (MINI).
* A Montgomery and Asberg Depression Rating Scale (MADRS) total score >=25 at the screening and baseline (day -1) visits and no more than a 5-point improvement from screening to baseline.

Exclusion Criteria:

* Treatment with DVS SR (Pristiq®) at any time in the past and/or venlafaxine, ie, Effexor® or Effexor XR®, 1 year prior to baseline.
* Treatment-resistant; eg, in the past 3 years if any of the following treatments have failed: (a) 3 or more previous adequate trials of >=2 classes of antidepressant medication, (b) electroconvulsive therapy, or (c) 2 adequate trials of psychotherapy (eg, behavior therapy, behavior-marital therapy).
* History or current evidence of gastrointestinal disease known to interfere with the absorption or excretion of drugs or a history of surgery known to interfere with the absorption or excretion of drugs.
* Known presence of raised intraocular pressure or history of narrow-angle glaucoma.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 439 (Actual)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (44):
- United States (44):
  - Birmingham Psychiatry Pharmaceutical Studies, Inc., Birmingham, Alabama
  - Arkansas Psychiatric Clinic Clinical Research Trials, P.A., Little Rock, Arkansas
  - Pacific Clinical Research Medical Group, Arcadia, California
  - Southwestern Research, Inc., Beverly Hills, California
  - Catalina Research Institute LLC, Chino, California
  - Pacific Clinical Research Medical Group, Orange, California
  - Pacific Clinical Research Medical Group, Upland, California
  - Western Affiliated Research Institute, Denver, Colorado
  - Radiant Research, Inc., Denver, Colorado
  - Connecticut Clinical Research, Cromwell, Connecticut
  - Comprehensive NeuroScience, Inc., St. Petersburg, Florida
  - Stedman Clinical Trials, LLC, Tampa, Florida
  - Janus Center for Psychiatric Research, West Palm Beach, Florida
  - Emory University Department of Psychiatry and Behavioral Sciences, Atlanta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Northwest Behavioral Research Center, Roswell, Georgia
  - Carman Research, Smyrna, Georgia
  - Capstone Clinical Research, Libertyville, Illinois
  - Deaconess Clinic Gateway Health Center Research Institute, Newburgh, Indiana
  - Via Christi Research, Witchita, Kansas
  - Westside Family Medical Center, P.C., Kalamazoo, Michigan
  - Radiant Research, Inc., Las Vegas, Nevada
  - Center For Emotional Fitness, Cherry Hill, New Jersey
  - Robert Wood Johnson Medical School, Piscataway, New Jersey
  - Social Psychiatry Research Institute, Brooklyn, New York
  - Medical & Behavioral Health Research PC, New York, New York
  - Metrolina Medical Research, Charlotte, North Carolina
  - Horizon Medical Services, PC, Bismarck, North Dakota
  - Legacy Pharma Research, Bismarck, North Dakota
  - North Coast Clinical Trials, Inc., Beechwood, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Summit Research Network (Oregon), Inc., Portland, Oregon
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Carolina Clinical Research Services, LLC, Columbia, South Carolina
  - Holston Medical Group, Bristol, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Bayou City Research, Ltd., Houston, Texas
  - Radiant Research, Inc., San Antonio, Texas
  - University of Virginia Health System Center for Psychiatric Clinical Research, Charlottesville, Virginia
  - Nelson Clinic, Richmond, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Summit Research Network (Seattle) LLC, Seattle, Washington
  - Independent Psychiatric Consultants, SC dba IPC Research, Waukesha, Wisconsin

REFERENCES:
- [Derived] Zilcha-Mano S, Wang X, Wajsbrot DB, Boucher M, Fine SA, Rutherford BR. Trajectories of Function and Symptom Change in Desvenlafaxine Clinical Trials: Toward Personalized Treatment for Depression. J Clin Psychopharmacol. 2021 Sep-Oct 01;41(5):579-584. doi: 10.1097/JCP.0000000000001435. PMID 34183490
- [Derived] Soares CN, Zhang M, Boucher M. Categorical improvement in functional impairment in depressed patients treated with desvenlafaxine. CNS Spectr. 2019 Jun;24(3):322-332. doi: 10.1017/S1092852917000633. Epub 2017 Nov 15. PMID 29140227
- [Derived] McIntyre RS, Fayyad R, Mackell JA, Boucher M. Effect of metabolic syndrome and thyroid hormone on efficacy of desvenlafaxine 50 and 100 mg/d in major depressive disorder. Curr Med Res Opin. 2016;32(3):587-99. doi: 10.1185/03007995.2015.1136603. Epub 2016 Jan 13. PMID 26709542
- [Derived] McIntyre RS, Fayyad RS, Guico-Pabia CJ, Boucher M. A Post Hoc Analysis of the Effect of Weight on Efficacy in Depressed Patients Treated With Desvenlafaxine 50 mg/d and 100 mg/d. Prim Care Companion CNS Disord. 2015 Jun 4;17(3):10.4088/PCC.14m01741. doi: 10.4088/PCC.14m01741. eCollection 2015. PMID 26644956
- [Derived] Kornstein SG, Clayton AH, Bao W, Guico-Pabia CJ. A pooled analysis of the efficacy of desvenlafaxine for the treatment of major depressive disorder in perimenopausal and postmenopausal women. J Womens Health (Larchmt). 2015 Apr;24(4):281-90. doi: 10.1089/jwh.2014.4900. PMID 25860107
- [Derived] Thase ME, Fayyad R, Cheng RF, Guico-Pabia CJ, Sporn J, Boucher M, Tourian KA. Effects of desvenlafaxine on blood pressure in patients treated for major depressive disorder: a pooled analysis. Curr Med Res Opin. 2015 Apr;31(4):809-20. doi: 10.1185/03007995.2015.1020365. Epub 2015 Mar 26. PMID 25758058
- [Derived] Soares CN, Endicott J, Boucher M, Fayyad RS, Guico-Pabia CJ. Predictors of functional response and remission with desvenlafaxine 50 mg/d in patients with major depressive disorder. CNS Spectr. 2014 Dec;19(6):519-27. doi: 10.1017/S1092852914000066. Epub 2014 Feb 26. PMID 24571916
- [Derived] Clayton AH, Kornstein SG, Dunlop BW, Focht K, Musgnung J, Ramey T, Bao W, Ninan PT. Efficacy and safety of desvenlafaxine 50 mg/d in a randomized, placebo-controlled study of perimenopausal and postmenopausal women with major depressive disorder. J Clin Psychiatry. 2013 Oct;74(10):1010-7. doi: 10.4088/JCP.12m08065. PMID 24229754
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3151A1-3364&StudyName=Study%20Evaluating%20Desvenlafaxine%20Succinate%20Sustained-Release%20%28DVS%20SR%29%20In%20The%20Treatment%20Of%20Peri-%20And%20Postmenopausal%20Women%20With%20Major%20De

RESULTS

PARTICIPANT FLOW:
Groups:
- Desvenlafaxine Succinate: Desvenlafaxine succinate sustained-release (DVS SR) 50 milligram tablets once daily for 10 weeks
- Placebo: Matching placebo tablets once daily for 10 weeks
Period: Overall Study
Arm/Group | Desvenlafaxine Succinate | Placebo
Started | 218 | 221
Treated | 217 | 217
Completed | 185 | 178
Not Completed | 33 | 43
Not completed — Adverse Event | 12 | 5
Not completed — Lack of Efficacy | 3 | 11
Not completed — Lost to Follow-up | 5 | 9
Not completed — Physician Decision | 0 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 8 | 7
Not completed — Discontinuation of study by sponsor | 0 | 1
Not completed — Other | 3 | 3
Not completed — Randomized, not treated | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Desvenlafaxine Succinate | Placebo | Total
Number analyzed (Participants) | 217 | 217 | 434
Age Continuous [Mean (Standard Deviation); unit: Years] | 53.1 (6.85) | 52.8 (6.58) | 53.0 (6.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 217 | 217 | 434
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hamilton Depression Scale (HAM-D17) at Week 8
Description: HAM-D17, clinician-rated interview, measures presence of depressive symptoms in 17 areas (symptoms such as depressed mood, guilty feelings, suicide, sleep disturbances, anxiety levels, & weight loss). Total score ranges from 0 to 52; higher scores indicate more severe depression. Change from baseline: score at observation minus score at baseline.
Time Frame: Baseline, Week 8
Population: Full Analysis Set (FAS) Population: randomized participants who had a baseline HAM-D17 score, took at least 1 dose of investigational product, and had at least 1 postbaseline HAM-D17 evaluation. Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Desvenlafaxine Succinate | Placebo
Number analyzed (Participants) | 216 | 216
Units on a scale
  Baseline | 22.8 (3.29) | 22.4 (3.51)
  Change at Week 8 | -9.7 (6.54) | -7.4 (6.74)
Statistical Analysis 1: Comparison: Desvenlafaxine Succinate vs Placebo; Null hypothesis: no difference between treatment groups; Test type: Superiority or Other; p = 0.004, ANCOVA — Analysis of Covariance used change from baseline at Week 8 as a response variable, site and treatment as factors, and baseline score as a covariate

2. Secondary Outcome: Number of Participants With Categorical Scores on Clinical Global Impression - Improvement (CGI-I)
Description: CGI-I: 7-point scale in which the clinician rated how much the participant's condition has changed compared to baseline. Scores ranged from 1 (very much improved) to 7 (very much worse). Improvement defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale. Higher score = more affected.
Time Frame: Week 8
Population: FAS; LOCF
Measure: Number; unit: participants
Arm/Group | Desvenlafaxine Succinate | Placebo
Number analyzed (Participants) | 216 | 216
participants
  Very Much Improved | 51 | 39
  Much Improved | 67 | 37
  Minimally Improved | 53 | 62
  No Change | 37 | 69
  Minimally Worse | 6 | 6
  Much Worse | 2 | 3
  Very Much Worse | 0 | 0
Statistical Analysis 1: Comparison: Desvenlafaxine Succinate vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — CGI-I analyzed as a categorical variable by Cochran-Mantel-Haenszel row-mean-score-difference test using ridit scores, controlling for the effect of region; p-value obtained from the alternative hypothesis of Row Mean Score Differences

3. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity (CGI-S) at Week 8
Description: CGI-S: 7-point clinician rated scale to assess severity of participant's current illness state; range: 1 (normal - not ill at all) to 7 (among the most extremely ill patients). Higher score = more affected. Change: score at observation minus score at baseline.
Time Frame: Baseline, Week 8
Population: FAS; LOCF
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Desvenlafaxine Succinate | Placebo
Number analyzed (Participants) | 216 | 216
Units on a scale
  Baseline | 4.4 (0.60) | 4.3 (0.53)
  Change at Week 8 | -1.5 (1.20) | -1.1 (1.24)
Statistical Analysis 1: Comparison: Desvenlafaxine Succinate vs Placebo; Test type: Superiority or Other; p = 0.002, ANCOVA — [p-value comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) - Total Score at Week 8
Description: Measures the overall severity of depressive symptoms. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). Change: score at observation minus score at baseline.
Time Frame: Baseline, Week 8
Population: FAS
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Desvenlafaxine Succinate | Placebo
Number analyzed (Participants) | 216 | 216
Units on a scale
  Baseline | 31.0 (3.76) | 30.6 (3.83)
  Change at Week 8 | -14.8 (9.09) | -11.6 (9.99)
Statistical Analysis 1: Comparison: Desvenlafaxine Succinate vs Placebo; Test type: Superiority or Other; p = 0.002, ANCOVA — [p-value comment as in outcome 1, analysis 1]

5. Secondary Outcome: Change From Baseline in Quick Inventory of Depressive Symptoms, 16 Question Self-report (QIDS-SR)
Description: This is a 16-item self reported questionnaire that measures depressive symptoms. Improvement reported as change in depressive score. Score ranges from 0 to 42, with higher numbers indicating more severe symptom reporting. Change: score at observation minus score at baseline.
Time Frame: Baseline, Week 8
Population: FAS; LOCF
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Desvenlafaxine Succinate | Placebo
Number analyzed (Participants) | 216 | 216
Units on a scale
  Baseline | 15.1 (3.22) | 14.8 (3.60)
  Change at Week 8 | -5.9 (4.93) | -5.2 (4.48)
Statistical Analysis 1: Comparison: Desvenlafaxine Succinate vs Placebo; Test type: Superiority or Other; p = 0.158, ANCOVA — [p-value comment as in outcome 1, analysis 1]

6. Secondary Outcome: Change From Baseline in Visual Analogue Scale for Pain (VAS-pain) at Week 8
Description: 10 centimeter (cm) line (Visual Analog Scale) marked by participant. Intensity of pain range (over past week): 0 = no pain to 10 = worst possible pain. Change: score at observation minus score at baseline.
Time Frame: Baseline, Week 8
Population: FAS; LOCF
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Desvenlafaxine Succinate | Placebo
Number analyzed (Participants) | 216 | 216
cm
  Baseline | 4.0 (2.90) | 4.0 (2.98)
  Change at Week 8 | -1.5 (2.69) | -0.8 (2.72)
Statistical Analysis 1: Comparison: Desvenlafaxine Succinate vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another participant, or 1 participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Desvenlafaxine Succinate | Placebo
Serious Adverse Events (participants affected / at risk) | 2/217 | 2/217
Other Adverse Events (participants affected / at risk) | 100/217 | 90/217
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Desvenlafaxine Succinate (N=217) | Placebo (N=217)
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Head Injury (Injury, poisoning and procedural complications) | 0 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 1 | 0
Subarachnoid Haemorrhage (Nervous system disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aneurysm Ruptured (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Desvenlafaxine Succinate (N=217) | Placebo (N=217)
Constipation (Gastrointestinal disorders) | 17 | 9
Diarrhoea (Gastrointestinal disorders) | 13 | 12
Dry Mouth (Gastrointestinal disorders) | 14 | 17
Nausea (Gastrointestinal disorders) | 24 | 16
Nasopharyngitis (Infections and infestations) | 15 | 12
Upper Respiratory Tract Infection (Infections and infestations) | 17 | 19
Dizziness (Nervous system disorders) | 14 | 10
Headache (Nervous system disorders) | 33 | 25

LIMITATIONS AND CAVEATS:
Baseline characteristics are available for all treated participants (434) and not all randomized participants (439).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.